CLINICAL TRIAL: NCT00784407
Title: Thyroid Surgery With the New Harmonic Scalpel: a Prospective Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hippocration General Hospital (Other)
Responsible Party: Department of Endocrine Surgery, 1st Department of Propaedeutic Surgery, Hippocratio General Hospital of Athens, Department of Endocrine Surgery, 1st Department of Propaedeutic Surgery, Hippocratio General Hospital of Athens, Athens Medical School, University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18858
Record Dates: First submitted 2008-11-03; First posted 2008-11-04 (Estimated); Last update posted 2008-11-04 (Estimated); Status verified 2008-10

CONDITIONS: Thyroidectomy
Keywords: thyroid surgery; total thyroidectomy; harmonic scalpel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOCUS (group A) (Active Comparator): Patients submitted to total thyroidectomy with the use of the FOCUS harmonic scalpel device
  Interventions: Device: harmonic scalpel device utilized intraoperatively
- HARMONIC ACE (group B) (Active Comparator): Patients submitted to total thyroidectomy with the use of the HARMONIC ACE harmonic scalpel device
  Interventions: Device: harmonic scalpel device utilized intraoperatively

INTERVENTIONS:
Device: harmonic scalpel device utilized intraoperatively — harmonic scalpel device utilized intraoperatively (FOCUS in group A and HARMONIC ACE in group B patients)

SUMMARY:
The objective of this study is to compare the results of total thyroidectomy using the new harmonic scalpel device (FOCUS) to that with the previously available harmonic scalpel device (HARMONIC ACE).

DETAILED DESCRIPTION:
Although the harmonic scalpel has been shown to be safe and effective in thyroid surgery, several surgeons consider the previously available instruments to be large and cumbersome, especially in terms of tissue fine grasping and dissection capabilities. To this context, an innovative technical improvement of the device for thyroid surgery has very recently been implemented and has been made available in 2008. Utilization of this new device, however, has not been evaluated in any study. The objective of this prospective randomized study is to compare the results of total thyroidectomy using the new harmonic scalpel device (FOCUS) to that with the previously available harmonic scalpel device (HARMONIC ACE) in respect to hemostasis, operative time and postoperative complications. All patients submitted to total thyroidectomy are randomized into two groups: those submitted to total thyroidectomy using the FOCUS device (group Α) and those with HARMONIC ACE (group Β).

ELIGIBILITY:
Inclusion Criteria:

* total thyroidectomy

Exclusion Criteria:

* hemithyroidectomy
* additional surgical procedures together with the total thyroidectomy (i.e. parathyroidectomy or cervical lymph node dissection)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-02; Primary Completion 2008-07 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Hemostasis | intraoperatively & postoperatively
Postoperative complications including laryngeal nerve palsy, hypocalcemia, hemorrhage, hematoma, wound infection and skin burn | postoperatively
Operative time | from skin incision to skin closure

SECONDARY OUTCOMES:
Length of hospital stay | postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Manouras, PhD, Principal Investigator — Department of Endocrine Surgery, 1st Department of Propaedeutic Surgery, Hippocratio General Hospital of Athens, Athens Medical School, University of Athens, Athens, Greece
Locations (1):
- Department of Endocrine Surgery, 1st Department of Propaedeutic Surgery, Hippocratio General Hospital of Athens, Athens Medical School, University of Athens, Athens, Abelokipoi (Q. Sofias 114 Av.), Greece